CLINICAL TRIAL: NCT04051879
Title: Influence of Reward and Punishment on Goal-directed and Habit Learning in Adolescent Anorexia Nervosa
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christina Wierenga, Associate Professor, University of California, San Diego
Other Study IDs: 182110
Record Dates: First submitted 2019-08-02; First posted 2019-08-09 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AN-R: Participants that meet Diagnostic And Statistical Manual Of Mental Disorders (DSM-V) criteria for Anorexia Nervosa restricting subtype.
- AN-BP: Participants that meet DSM-V criteria for Anorexia Nervosa binging/purging subtype.
- Healthy Controls: Participants that do not meet DSM-V criteria for any disorder.

SUMMARY:
The proposed study of adolescents with anorexia nervosa (AN) will examine the association of behavioral differences in constructs of decision making, brain structure and connectivity, and eating disorder (ED) symptoms. This study tests the novel hypothesis that goal-directed and habit learning for reward and punishment is altered in AN and is uniquely associated with divergent symptoms and differences in corticostriatal connectivity and microstructural integrity. We will recruit 78 females currently ill with AN and 26 controls ages 13-17 to investigate how goal-directed and habit learning for reward and punishment correspond to 1) clinical symptoms collected via interviews, self-report assessments, and ecological momentary assessment (EMA), and 2) brain structure and connectivity in the resting state. Data collection will rely on a technology called functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

AN Group:

* Between the ages of 13 and 17 years old
* Meet DSM-V criteria for AN-R or AN-BP
* Medically stable per American Academy of Pediatrics and the Society of Adolescent Medicine requirements, at least 75% adjusted ideal body weight, but still symptomatic as assessed by the Eating Disorders Examination and clinical report
* Be at least 75% of adjusted ideal body weight

Healthy Control Group:

* Between the ages of 13 and 17 years old

Exclusion Criteria:

All Groups:

* Psychotic illness/other mental illness requiring hospitalization
* Current dependence on drugs or alcohol defined by DSM IV criteria. Additionally, positive test results for drug use on the day of the scan, apart of marijuana, will result in cancelling or rescheduling the scan because acute use will impact MRI measures.
* Physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight
* Neurological disorder, neurodevelopmental disorder, or history of head injury with >30 min loss of consciousness
* Any contraindication to undergoing an MRI
* Primary obsessive compulsive disorder or primary major depressive disorder

Additional Exclusion Criteria for AN Group:

* If taking other psychotropic medication, any change in dosage in the 2 weeks before scanning

Additional Exclusion Criteria for Healthy Control Group:

* Meet or met criteria for the diagnosis of any psychiatric disorder in their lifetime
* Any history of binge eating or purging behaviors, including self-induced vomiting, laxative or diuretic misuse
* Use of any psychoactive or other medication known to affect mood or concentration in the last 3 months
* Have maintained 90% to 120% ideal body weight since menarche

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will recruit from a clinical sample for the AN groups. We will recruit from a community sample for the healthy control group.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Learning Task | Computer Task (Baseline)
  A learning computer task will be used to dissociate model-based and model-free learning.
Brain Function | fMRI Scan (Baseline)
  Functional Magnetic Resonance Imaging will be used to correlate brain function with a weighting factor (ω), representing the relative balance between learning biases.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wierenga, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided